CLINICAL TRIAL: NCT00766090
Title: A Multi-Centre, Randomized, Double Blind Cross-over Study to Assess the Non-inferiority of GW685698X 200mcg Once Daily and 100mcg Twice Daily in Adult and Adolescent Patients With Asthma
Brief Title: Safety and Efficacy of GW685698X an Inhaled Corticosteroid Once Daily and Twice Daily for the Treatment of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112202
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GW685698X (Experimental)
  Interventions: Drug: GW685698X

INTERVENTIONS:
Drug: GW685698X — Inhaled Corticosteroid

SUMMARY:
The purpose of this study is to compare once and twice daily GW685698 in asthma

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of Asthma
* Reversibility ≥ 12% and ≥200mls reversibility of FEV1 within approximately 30-minutes following 2 to 4 puffs of albuterol
* FEV1 between 40-85% predicted
* Currently on short acting beta2 agonist therapy

Key Exclusion Criteria:

* History of life threatening asthma
* Respiratory Infection or oropharyngeal candidiasis
* Asthma exacerbation
* Uncontrolled disease or clinical abnormality
* Allergies
* Taking another Investigational medications or other prohibited medications

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (15):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Woodcock A, Bleecker ER, Busse WW, Lotvall J, Snowise NG, Frith L, Jacques L, Haumann B, Bateman ED. Fluticasone furoate: once-daily evening treatment versus twice-daily treatment in moderate asthma. Respir Res. 2011 Dec 21;12(1):160. doi: 10.1186/1465-9921-12-160. PMID 22188590
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112202 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants (par.) at screening entered a 14-day Run-in Period. Par. were then randomized to 1 of 12 sequences: 6 had placebo and two doses of fluticasone furoate (FF), and 6 had placebo and two doses of fluticasone proprionate (FP) (allocation ratio of 7:2 [FF:FP]). 320 par. were screened and 190 were randomized.
Groups:
- Sequence 1: Placebo, FF 200 µg, FF 100 µg: Participants received placebo twice daily (BID), fluticasone furoate (FF) 200 microgram (µg) inhalation powder once daily (OD) in the evening, and FF 100 µg inhalation powder twice daily (BID) in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 2: Placebo, FF 100 µg, FF 200 µg: Participants received placebo BID, FF 100 µg inhalation powder BID, and FF 200 µg inhalation powder OD in the evening in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 3: FF 100 µg, Placebo, FF 200 µg: Participants received FF 100 µg inhalation powder BID, placebo BID, and FF 200 µg inhalation powder OD in the evening in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 4: FF 100 µg, FF 200 µg, Placebo: Participants received FF 100 µg inhalation powder BID, FF 200 µg inhalation powder OD in the evening, and placebo BID in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 5: FF 200 µg, Placebo, FF 100 µg: Participants received FF 200 µg inhalation powder OD in the evening, placebo BID, and FF 100 µg inhalation powder BID in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 6: FF 200 µg, FF 100 µg, Placebo: Participants received FF 200 µg inhalation powder OD in the evening, FF 100 µg inhalation powder BID, and placebo BID in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 7: Placebo, FP 200 µg, FP 100 µg: Participants received placebo twice daily (BID), fluticasone propionate (FP) 200 microgram (µg) inhalation powder once daily (OD) in the evening, and FP 100 µg inhalation powder twice daily (BID) in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a DISKUS inhaler for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 8: Placebo, FP 100 µg, FP 200 µg: Participants received placebo BID, FP 100 µg inhalation powder BID, and FP 200 µg inhalation powder OD in the evening in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a DISKUS inhaler for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 9: FP 100 µg, Placebo, FP 200 µg: Participants received FP 100 µg inhalation powder BID, placebo BID, and FP 200 µg inhalation powder OD in the evening in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a DISKUS inhaler for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 10: FP 100 µg, FP 200 µg, Placebo: Participants received FP 100 µg inhalation powder BID, FP 200 µg inhalation powder OD in the evening, and placebo BID in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a DISKUS inhaler for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 11: FP 200 µg, Placebo, FP 100 µg: Participants received FP 200 µg inhalation powder OD in the evening, placebo BID, and FP 100 µg inhalation powder BID in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a DISKUS inhaler for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Sequence 12: FP 200 µg, FP 100 µg, Placebo: Participants received FP 200 µg inhalation powder OD in the evening, FP 100 µg inhalation powder BID, and placebo BID in Treatment Periods 1, 2, and 3, respectively. All treatments were administered via a DISKUS inhaler for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
Period: Treatment Period 1 (28 Days)
Arm/Group | Sequence 1: Placebo, FF 200 µg, FF 100 µg | Sequence 2: Placebo, FF 100 µg, FF 200 µg | Sequence 3: FF 100 µg, Placebo, FF 200 µg | Sequence 4: FF 100 µg, FF 200 µg, Placebo | Sequence 5: FF 200 µg, Placebo, FF 100 µg | Sequence 6: FF 200 µg, FF 100 µg, Placebo | Sequence 7: Placebo, FP 200 µg, FP 100 µg | Sequence 8: Placebo, FP 100 µg, FP 200 µg | Sequence 9: FP 100 µg, Placebo, FP 200 µg | Sequence 10: FP 100 µg, FP 200 µg, Placebo | Sequence 11: FP 200 µg, Placebo, FP 100 µg | Sequence 12: FP 200 µg, FP 100 µg, Placebo
Started | 25 | 27 | 23 | 26 | 23 | 23 | 6 | 8 | 7 | 8 | 7 | 7
Completed | 22 | 27 | 23 | 25 | 23 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Not Completed | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (14 Days)
Arm/Group | Sequence 1: Placebo, FF 200 µg, FF 100 µg | Sequence 2: Placebo, FF 100 µg, FF 200 µg | Sequence 3: FF 100 µg, Placebo, FF 200 µg | Sequence 4: FF 100 µg, FF 200 µg, Placebo | Sequence 5: FF 200 µg, Placebo, FF 100 µg | Sequence 6: FF 200 µg, FF 100 µg, Placebo | Sequence 7: Placebo, FP 200 µg, FP 100 µg | Sequence 8: Placebo, FP 100 µg, FP 200 µg | Sequence 9: FP 100 µg, Placebo, FP 200 µg | Sequence 10: FP 100 µg, FP 200 µg, Placebo | Sequence 11: FP 200 µg, Placebo, FP 100 µg | Sequence 12: FP 200 µg, FP 100 µg, Placebo
Started | 22 | 27 | 23 | 25 | 23 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Completed | 22 | 27 | 22 | 25 | 23 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (28 Days)
Arm/Group | Sequence 1: Placebo, FF 200 µg, FF 100 µg | Sequence 2: Placebo, FF 100 µg, FF 200 µg | Sequence 3: FF 100 µg, Placebo, FF 200 µg | Sequence 4: FF 100 µg, FF 200 µg, Placebo | Sequence 5: FF 200 µg, Placebo, FF 100 µg | Sequence 6: FF 200 µg, FF 100 µg, Placebo | Sequence 7: Placebo, FP 200 µg, FP 100 µg | Sequence 8: Placebo, FP 100 µg, FP 200 µg | Sequence 9: FP 100 µg, Placebo, FP 200 µg | Sequence 10: FP 100 µg, FP 200 µg, Placebo | Sequence 11: FP 200 µg, Placebo, FP 100 µg | Sequence 12: FP 200 µg, FP 100 µg, Placebo
Started | 22 | 27 | 22 | 25 | 23 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Completed | 22 | 27 | 21 | 25 | 21 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Not Completed | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (14 Days)
Arm/Group | Sequence 1: Placebo, FF 200 µg, FF 100 µg | Sequence 2: Placebo, FF 100 µg, FF 200 µg | Sequence 3: FF 100 µg, Placebo, FF 200 µg | Sequence 4: FF 100 µg, FF 200 µg, Placebo | Sequence 5: FF 200 µg, Placebo, FF 100 µg | Sequence 6: FF 200 µg, FF 100 µg, Placebo | Sequence 7: Placebo, FP 200 µg, FP 100 µg | Sequence 8: Placebo, FP 100 µg, FP 200 µg | Sequence 9: FP 100 µg, Placebo, FP 200 µg | Sequence 10: FP 100 µg, FP 200 µg, Placebo | Sequence 11: FP 200 µg, Placebo, FP 100 µg | Sequence 12: FP 200 µg, FP 100 µg, Placebo
Started | 22 | 27 | 21 | 25 | 21 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Completed | 22 | 27 | 20 | 25 | 21 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (28 Days)
Arm/Group | Sequence 1: Placebo, FF 200 µg, FF 100 µg | Sequence 2: Placebo, FF 100 µg, FF 200 µg | Sequence 3: FF 100 µg, Placebo, FF 200 µg | Sequence 4: FF 100 µg, FF 200 µg, Placebo | Sequence 5: FF 200 µg, Placebo, FF 100 µg | Sequence 6: FF 200 µg, FF 100 µg, Placebo | Sequence 7: Placebo, FP 200 µg, FP 100 µg | Sequence 8: Placebo, FP 100 µg, FP 200 µg | Sequence 9: FP 100 µg, Placebo, FP 200 µg | Sequence 10: FP 100 µg, FP 200 µg, Placebo | Sequence 11: FP 200 µg, Placebo, FP 100 µg | Sequence 12: FP 200 µg, FP 100 µg, Placebo
Started | 22 | 27 | 20 | 25 | 21 | 23 | 6 | 8 | 6 | 8 | 7 | 7
Completed | 22 | 26 | 20 | 24 | 20 | 22 | 6 | 8 | 6 | 8 | 7 | 6
Not Completed | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FF 200 µg, FF 100 µg, and Placebo Via DPI: Participants received FF 200 µg inhalation powder OD in the evening, FF 100 µg inhalation powder BID, and placebo BID in one of the three treatment periods. All treatments were administered via a Dry Powder Inhaler (DPI) for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- FP 200 µg, FP 100 µg, and Placebo Via DISKUS: Participants received FP 200 µg inhalation powder OD in the evening, FP 100 µg inhalation powder BID, and placebo BID in one of the three treatment periods. All treatments were administered via a DISKUS for 28 days. Each of the 3 treatment periods was separated by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- Total: Total of all reporting groups
Arm/Group | FF 200 µg, FF 100 µg, and Placebo Via DPI | FP 200 µg, FP 100 µg, and Placebo Via DISKUS | Total
Number analyzed (Participants) | 147 | 43 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (15.30) | 35.2 (16.03) | 32.3 (15.51)
Gender [Count of Participants; unit: Participants]
  Female | 87 | 21 | 108
  Male | 60 | 22 | 82
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage (HER) | 50 | 20 | 70
  American Indian (AI) or Alaska Native (AN) | 1 | 0 | 1
  Japanese/East Asian HER/South East Asian HER | 2 | 1 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 90 | 22 | 112
  African American/African HER & AI or AN & White | 1 | 0 | 1
  African American/African Heritage & White | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) at Day 28 of the Relevant Treatment Period
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured electronically by spirometry. Trough FEV1 was the evening pre-dose, pre-rescue bronchodilator FEV1 measurement taken on Day 28 of the relevant treatment period. The analysis was performed using mixed model analysis of covarience (ANCOVA) with fixed effects of treatment, period, sex, and age. Participants were fitted as a random effect, and the period Baseline measurement was included as part of a bivariate response.
Time Frame: Day 28 of the relevant treatment period (up to Study Day 112)
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Participants received placebo BID via the Dry Powder Inhaler (DPI) or the DISKUS inhaler for 28 days during one of the 3 treatment periods. Each treatment period was followed by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- FF 200 µg OD: Participants received FF 200 µg inhalation powder OD in the evening from the DPI for 28 days during one of the 3 treatment periods. Each treatment period was followed by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- FF 100 µg BID: Participants received FF 100 µg inhalation powder BID from the DPI for 28 days during one of the 3 treatment periods. Each treatment period was followed by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- FP 200 µg OD: Participants received FP 200 µg inhalation powder OD PM from the DISKUS inhaler for 28 days during one of the 3 treatment periods. Each treatment period was followed by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
- FP 100 µg BID: Participants received FP 100 µg inhalation powder BID from the DISKUS inhaler for 28 days during one of the 3 treatment periods. Each treatment period was followed by a washout period of 14 days. Participants were provided supplemental albuterol/salbutamol (inhalation aerosol) to be used as needed throughout the study.
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 187 | 140 | 142 | 42 | 43
Liters | 2.605 (0.0434) | 2.714 (0.0444) | 2.703 (0.0443) | 2.693 (0.0535) | 2.737 (0.0533)
Statistical Analysis 1: Comparison: Placebo vs FF 200 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.108, 95% CI 2-sided [0.064 to 0.153]
Statistical Analysis 2: Comparison: Placebo vs FF 100 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [0.054 to 0.142]
Statistical Analysis 3: Comparison: Placebo vs FP 200 µg OD; Test type: Superiority or Other; p = 0.020, ANCOVA; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.014 to 0.161]
Statistical Analysis 4: Comparison: FF 200 µg OD vs FF 100 µg BID; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the lower limit of the confidence interval (0.025, 1-sided significance level) for the mean difference in trough FEV1 of FF 200 µg OD versus FF 100 µg BID was greater than -110 milliliters; p = 0.641, ANCOVA; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.035 to 0.056]
Statistical Analysis 5: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.132, 95% CI 2-sided [0.059 to 0.205]

2. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE) Throughout the Three 28-day Treatment Periods
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations. Refer to the general AE/SAE module for a list of AEs (occuring at a frequency threshold >=3%) and SAEs.
Time Frame: From the first dose of the study medication up to Week 16/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 187 | 140 | 142 | 42 | 43
participants
  Any AE | 26 | 22 | 26 | 2 | 3
  Any SAE | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: 24-hour Urinary Cortisol Excretion at Day 28 of the Relevant Treatment Period
Description: A 24-hour urine sample was collected, and the 24-hour urinary cortisol excretion was analyzed at Day 28 of the relevant treatment period.
Time Frame: Day 28 of the relevant treatment period (up to Study Day 112)
Population: Urine Cortisol (UC) Population: participants who had both a Baseline urine sample and at least one urine sample from the end of a treatment period that did not have confounding factors that could affect the interpretation of results
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per 24 hours
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 153 | 118 | 116 | 35 | 39
Nanomoles per 24 hours | 53.94 (66.423) | 40.25 (92.316) | 45.13 (87.181) | 56.16 (94.259) | 47.56 (84.896)

4. Secondary Outcome: Number of Participants With Evidence of Oropharyngeal Candidiasis at Day 0 and Day 28 of the Relevant Treatment Period
Description: Detailed oropharyngeal examination for visual evidence of oropharyngeal candidiasis was performed at Day 0 (clinic visits 2, 4, and 6) and Day 28 (clinic visits 3, 5, and 7) of the relevant treatment period.
Time Frame: Day 0 and Day 28 of the relevant treatment period (up to Study Day 112)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 187 | 140 | 142 | 42 | 43
participants
  Day 0: Yes, n=187, 140, 142, 42, 43 | 0 | 0 | 0 | 0 | 0
  Day 0: No, n=187, 140, 142, 42, 43 | 187 | 140 | 142 | 42 | 43
  Day 28: Yes, n=178, 139, 140, 42, 42 | 0 | 0 | 0 | 0 | 0
  Day 28: No, n=178, 139, 140, 42, 42 | 178 | 139 | 140 | 42 | 42

5. Secondary Outcome: Systolic and Diastolic Blood Pressure at Day 0 and Day 28 of the Relevant Treatment Period
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured at Day 0 (clinic visits 2, 4, and 6) and Day 28 (clinic visits 3, 5, and 7) of the relevant treatment period.
Time Frame: Day 0 and Day 28 of the relevant treatment period (up to Study Day 112)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 187 | 140 | 142 | 42 | 43
millimeters of mercury (mmHg)
  SBP: Day 0, n=187, 140, 142, 42, 43 | 120.1 (12.08) | 118.3 (11.96) | 119.5 (12.28) | 122.1 (13.55) | 121.3 (12.10)
  SBP: Day 28, n=178, 139, 140, 42, 42 | 119.6 (12.76) | 120.5 (13.31) | 120.6 (12.71) | 120.4 (11.92) | 120.1 (10.58)
  DBP: Day 0, n=187, 140, 142, 42, 43 | 75.8 (8.26) | 74.6 (7.69) | 76.0 (8.03) | 77.5 (9.98) | 76.6 (8.73)
  DBP: Day 28, n=178, 139, 140, 42, 42 | 75.8 (8.45) | 74.9 (8.12) | 76.4 (7.97) | 76.0 (7.81) | 75.7 (8.90)

6. Secondary Outcome: Heart Rate at Day 0 and Day 28 of the Relevant Treatment Period
Description: Heart rate was measured at Day 0 (clinic visits 2, 4, and 6) and Day 28 (clinic visits 3, 5, and 7) of the relevant treatment period.
Time Frame: Day 0 and Day 28 of the relevant treatment period (up to Study Day 112)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Number analyzed (Participants) | 187 | 140 | 142 | 42 | 43
beats per minute
  Day 0, n=187, 140, 142, 42, 43 | 77.0 (9.53) | 76.4 (9.27) | 77.6 (8.71) | 74.5 (9.22) | 75.8 (8.12)
  Day 28, n=178, 139, 140, 42, 42 | 76.6 (8.79) | 76.9 (9.32) | 77.7 (9.47) | 74.7 (7.96) | 74.6 (8.49)

7. Secondary Outcome: Number of Participants Who Withdrew Due to Worsening of Asthma During the Three Treatment Periods
Description: Participants were withdrawn from the study due to worsening of asthma (lack of efficacy) if they experienced a clinical asthma exacerbation or if clinic FEV1 fell below the FEV1 stability limit, or if during the 7 days immediately preceeding a visit the participant experienced either four or more days in which the PEF had fallen below the PEF stability limit or three or more days in which >=12 inhalations/day of albuterol/salbutamol were used. A clinical asthma exacerbation is defined as the worsening of asthma requiring emergency room visits, hospitalization, or treatment with an asthma medication (inhaled or systemic corticosteroids) other than study medication or rescue salbutamol/albuterol.
Time Frame: From the first dose of the study medication up to Week 16/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | FF 200 µg, FF 100 µg, and Placebo Via DPI | FP 200 µg, FP 100 µg, and Placebo Via DISKUS
Number analyzed (Participants) | 147 | 43
participants | 5 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of the study medication up to Week 16/Early Withdrawal.
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | Placebo | FF 200 µg OD | FF 100 µg BID | FP 200 µg OD | FP 100 µg BID
Serious Adverse Events (participants affected / at risk) | 0/187 | 0/140 | 0/142 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 2/187 | 7/140 | 7/142 | 0/42 | 0/43
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=187) | FF 200 µg OD (N=140) | FF 100 µg BID (N=142) | FP 200 µg OD (N=42) | FP 100 µg BID (N=43)
Upper respiratory tract infection (Infections and infestations) | 2 | 7 | 7 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.